CLINICAL TRIAL: NCT05531916
Title: Compression Therapy as a Prophylactic Method Against Paclitaxel-induced Peripheral Neuropathy: a Prospective Self-controlled Trial
Brief Title: Compression Therapy as a Prophylactic Method Against CIPN: a Prospective Self-controlled Trial
Acronym: CIPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Chunyan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2022-306-01
Record Dates: First submitted 2022-08-27; First posted 2022-09-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Nasopharyngeal Carcinoma; CIPN - Chemotherapy-Induced Peripheral Neuropathy
Keywords: Paclitaxel; Compression therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: The Account and IWRS end of the clinical trial randomization system of Sun Yat-sen University Cancer Center (SYSUCC) randomly determined the limb (left or right) of the participants to receive intervention, and the hand and foot on the same side were classified into the same group during the randomization process.
Who Masked: Outcomes Assessor
Masking Description: Evaluator blind design was adopted, and all evaluations were made after the participants had received the intervention and withdrawn the intervention. At this time, the blinded evaluator did not know the tribal groups, while both the participants and researchers knew the trial groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants wear pressurized gloves and foot caps for 15 minutes before their chemotherapy treatment, during the treatment, and for 15 minutes after it ended.
  Interventions: Other: Pressurized gloves and foot caps
- Group B (No Intervention): No intervention was done before and after chemotherapy with paclitaxels.

INTERVENTIONS:
Other: Pressurized gloves and foot caps — Using pressurized gloves and foot caps in order to prevent chemotherapy-induced peripheral neuropathy (CIPN).
  Arms: Group A

SUMMARY:
This is a single-center, self-controlled, evaluator-blinded prospective study, which applies pressurized gloves and foot caps to prevent paclitaxel-induced peripheral neuropathy in patients with nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 70
* ECOG physical status score: 0-2
* Newly diagnosed patients who have not received antitumor therapy
* Nasopharyngeal carcinoma confirmed by pathology
* Paclitaxel is included in the chemotherapy regimen
* Laboratory examination results within one week before enrollment should meet the following conditions: neutrophils (ANC) ≥1.5×109/L, platelets (PLT) ≥80×109/L, total bilirubin (TBI) ≤1.5× upper limit of normal value (2mg/ dL), ALT and AST ≤2× upper limit of normal value
* Patients voluntarily participate and provide written informed consent

Exclusion Criteria:

* Patients with peripheral neuropathy, hand-foot syndrome, and dermatomyositis
* Patients with missing fingers or toes
* Patients with Raynaud's syndrome and peripheral vascular ischemia
* Pregnant or lactating women
* Those considered unsuitable for inclusion by the researcher

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation change in CTCAE 5.0 grade for CIPN (The most severe grade is the final grade) | Pretreatment (baseline=0), just after 15 minutes of each treatment cycle (each cycle of chemotherapy is 21 days) , 3 and 6 months after chemotherapy completion.
  The incidence of common adverse event evaluation criteria (CTCAE) 5.0 ≥ 2°CIPN after compression therapy with pressurized gloves and foot caps is used to objectively assess the peripheral neurotoxicity of chemotherapy. The grade of CTCAE 5.0 CIPN before treatment was the baseline (=0). We assess changes from baseline at 15 minutes after the end of each cycle, 3 and 6 months after the end of treatment. (The duration of chemotherapy varies according to the type of paclitaxel and the interval of each cycle of chemotherapy is 21 days). CIPN includes the symptoms of a sensory nerve and motor nerve injury. The symptoms are graded from 1 to 5, indicating none, mild, severe, life-threatening, and death. The higher the grade, the worse the neurotoxicity. The most severe grade is the final grade for each patient.

SECONDARY OUTCOMES:
EORTC QLQ-CIPN20 score | Pretreatment (baseline), just after 15 minutes of each treatment cycle (each cycle of chemotherapy is 21 days) , 3 and 6 months after chemotherapy completion.
  The European Organization for Research and Treatment of Cancer Evaluation Scale of Chemotherapy-Induced Peripheral Neuropathy (EORTC QLQ-CIPN20) is a validated tool to objectively assess the peripheral neurotoxicity of chemotherapy. The evaluation was performed before treatment, 15 minutes after each cycle of chemotherapy, and 3 and 6 months after the end of treatment. This scale includes the symptoms of sensory nerve, motor nerve, and autonomic nerve injury and its impact on life. A total of 20 items are included. Each item is graded from 1 to 4, indicating none, occasionally, often, and very often. According to the patient's self-reported score, the higher the score, the worse the quality of life.
EORTC QLQ-C30 score | Pretreatment (baseline), just after 15 minutes of each treatment cycle (each cycle of chemotherapy is 21 days), 3 and 6 months after chemotherapy completion.
  The European Organization for Cancer Research and Treatment QLQ-C30 （EORTC QLQ-C30）: a quality of life instrument for use in international clinical trials in oncology. The evaluation was performed before treatment, 15 minutes after each cycle of chemotherapy, and 3 and 6 months after the end of treatment. A total of 30 items are included. Each item is graded from 1 to 4, except for items 29 and 30, indicating not at all, a little, quite a bit, and very much, with higher scores indicating poorer quality of life.
NRS score | Pretreatment（baseline), just after 15 minutes of each treatment cycle (each cycle of chemotherapy is 21 days.)
  The Numerical Rating Scale (NRS) scale is a validated tool to objectively assess the tolerance of participants for gloves and coats, with a minimum score of 0 and a maximum of 10. A score of 0 indicates complete tolerance, a score of 1-3 indicates mild intolerance, a score of 4-6 indicates moderate intolerance, and a score of 7-10 indicates severe intolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No